CLINICAL TRIAL: NCT00479609
Title: A Randomised Placebo Controlled Study of Transdermal Testosterone Therapy to Investigate the Efficacy and Safety in Men With Abdominal Obesity, Low Testosterone Levels and Early Stages of the Metabolic Cluster Syndrome.
Brief Title: Testosterone Therapy in Men With Low Testosterone Levels and Metabolic Syndrome or Early Stages of Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Southern Hospital Stockholm (Unknown); UroHealth Skövde (Unknown); Universitätsklinikum MünsterInstitut für Reproduktionsmedizin (Unknown); Krankenanstalt der Stadt Wien Rudolfstiftung (Unknown); Medical University of Graz (Other); Krankenhaus der Stadt Wien Lainz (Unknown); Medical University of Vienna (Other); Endokrinologikum Hamburg (Unknown); Charite University, Berlin, Germany (Other)
Responsible Party: Stefan Arver Associate Prof, Sr Physician, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARTinMMS
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Metabolic Syndrome
Keywords: Insulin resistance; Glucose tolerance; Type 2 diabetes; Androgen sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo gel
  Interventions: Drug: Placebo
- 2 (Active Comparator): Transdermal testostrone therapy
  Interventions: Drug: Transdermal testosterone therapy

INTERVENTIONS:
Drug: Transdermal testosterone therapy — testosterone 1% hydroalcohol gel
  Arms: 2
Drug: Placebo — Placebo gel
  Arms: 1

SUMMARY:
Men with metabolic syndrome often have lower than normal testosterone levels and low testosterone levels have been suggested to predispose for development of type2 diabetes. The aim of the study is to evaluate if normalisation of serum testosterone levels in men with metabolic syndrome (Abdominal obesity, hypertension, dyslipidemia, insulin resistance and pre-diabetes or overt type diabetes)improves sensitivity to insulin and improves the signs of the metabolic syndrome

DETAILED DESCRIPTION:
Background The metabolic syndrome constitutes a cluster of risk factors for cardiovascular disease with increased morbidity and mortality. In essence the metabolic syndrome is referred to as a concomitant occurrence of hypertension, hyperlipidemia, impaired glucose tolerance with insulin resistance and abdominal obesity. The presence of abdominal obesity seems to be a key factor in development of the metabolic derangements that occur and is a part of all different definitions that are currently used as diagnostic criteria's for the metabolic syndrome. A number of studies have verified a serious prognosis for males (and females) presenting with the abdominal obesity.

The term metabolic syndrome alludes to a common mechanism behind the development of the different sings of this condition but so far the etiological interrelationship is not known. In males with the metabolic syndrome low serum testosterone levels is a common finding and data from some longitudinal studies suggest that low testosterone levels precedes the development of abdominal obesity and seem to facilitate later development of hypertension, hyperlipidemia and hyperglycemia. A few smaller studies have tested the hypothesis that testosterone therapy may have a beneficial metabolic effect in males with the metabolic syndrome and implicated that low testosterone levels is a part of disease facilitating factors in these males.

Current study The current study "ARTinMMS" is an interventional phase IV study in males (30-70 years inclusive) with early stages of the metabolic syndrome defined as abdominal obesity, glucose intolerance or overt type 2 diabetes defined according to the criteria's suggested by the International Federation for Diabetes. The study is a 24 weeks randomized placebo controlled parallel group multi-centre study where males with serum testosterone levels below 12 nmol/L will be treated with testosterone/placebo (total duration of study including follow-up visit 26-27 weeks). The primary endpoint of the study is assessment of insulin sensitivity by measurement of fasting plasma glucose and insulin levels and calculated according to the QUICKI formula. In addition glucose tolerance will be tested with a standard oral glucose tolerance test as well as assessment of blood lipids and blood pressure.

A total of 176 males will be recruited and randomized for the study after a screening procedure to verify eligibility for the study. Males who can participate must fulfil a series of inclusion and exclusion criteria, which in addition to the metabolic syndrome and low testosterone levels require HbA1c levels below 7,5%, stable blood pressure control and cholesterol levels below 8 mmol/L. Medical treatment for these conditions are accepted but diabetes treatment is limited to metformin.

Before entering into the study and during the study males will be followed with blood tests and glucose tolerance assessment and physical examination. In all the study requires five clinical visits, Base-line observations and randomization visit, two visits during the treatment phase (after 12 and 23 weeks of therapy) and a follow-up visit after cessation of therapy.

A few exploratory variables will be assess such as markers for changes in cholesterol metabolism, adiponectin and all subjects in the study will be characterized with genotype analysis of CAG repeat polymorphism of the androgen receptor. A subset of patients will be examined with CT of the abdomen to assess eventual changes in intra abdominal fat mass and liver attenuation.

Safety procedures involve assessment of the prostate (digital rectal examination and PSA levels) and Hb levels at baseline and throughout the study.

Study medication Males enrolled in the study will be treated with daily application of 7,5 g of a 1% testosterone hydroalcoholic gel (75 mg of testosterone applied on specified skin sites) or a placebo gel.

Time plan The study is planned to start in q2 2007 at 12 different centres, in Austria, Germany and Sweden. Each centre is anticipated to recruit 10 -30 subjects during a 2 months period. To facilitate recruitment newspaper advertising and web based eligibility screening will be used if feasible. After an 1-3 weeks screening period eligible subjects are randomized to active or placebo therapy. Two evaluations are made during the treatment phase the first after 12 and the second after 24 weeks. Efficacy and safety assessments are performed at these visits. Competitive enrolment is used after the first six weeks of the recruitment period enabling all centres to recruit an up-front agreed number of subjects.

Data capturing and laboratory routines A centralized internet based system will be used for data capturing, communication with the study staff and automatic entry of laboratory data. All laboratory analysis will be performed at or through a core laboratory (LFK in Kiel). A paper CRF will be used for primary entry of patient data which are subsequently transcribed into an electronic CRF. All study centres will be trained during the investigators meeting in management of the data capturing system

ELIGIBILITY:
Inclusion Criteria:

1. Male 30 to 70 years (inclusive)
2. Metabolic syndrome defined according to the International Diabetes Foundation (IDF):

   1. Abdominal obesity (waist circumference > 94 cm for European men) and any two of the following criteria
   2. Triglycerides > 1.7 mmol/L or specific treatment for this
   3. HDL < 1.03 nmol/L or specific therapy for this
   4. Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg or treatment for this.
   5. Fasting plasma glucose ≥ 5.6 mmol/L (venous glucose ≥ 6.1 mmol/L) or previously diagnosed type 2 diabetes mellitus defined by: Fasting plasma glucose ≥ 7.8 mmol/L on two occasions, or random glucose ≥ 11.1 mmol/L and classic symptoms of type 2 diabetes
3. Impaired glucose tolerance If the definition of the metabolic syndrome, as described above, is fulfilled but fasting plasma glucose ≤ 5.6 mmol/L (fasting venous glucose is < 6.1 mmol/L) the result of an oral glucose tolerance test must be classified as reduced glucose tolerance with a venous blood glucose 7.8 - 11.1 mmol/L or higher 120 min after intake of 75 g of glucose in a water solution (2h OGTT) (www.diabetes.org/main/info/pre-diabetes.jsp)
4. Hypogonadism, S-Testosterone <12 nmol/L taken at 7:00-10:00 a.m. Sample taken less than 2 months before inclusion in the study.
5. Screening value of HbA1c <7.5 %
6. Weight < 110 kg
7. Body Mass Index (BMI) < 35
8. Hematocrit < 50%
9. Signed Written informed consent obtained -

Exclusion Criteria:

1. Ongoing pharmacological treatment of type 2 diabetes except for metformin.
2. Use of androgen therapy or anabolic steroids within 6 months of entry into the study.
3. Known congestive heart failure, progressing angina pectoris or a history of myocardial infarction within the last 12 months.
4. Known untreated pituitary disease.
5. A history of significant renal or liver disease or any malignancy.
6. Use of drugs interfering with androgens; spironolactone, Ketoconazol, corticosteroids, cimetidine, fentiazines, tricyclic antidepressants, anabolic steroids, 5-alfa reductase inhibitors, antiestrogens.
7. Prostate Specific Antigen (PSA) > 4 ng/ml.
8. Suspected malignancy after prostata palpation, unless biopsy shows the opposite.
9. Malignant tumour of the mammary gland
10. Ongoing micturition problem severely affecting patient's daily living as judged by the investigator.
11. Any contraindication for treatment with testosterone 1% hydroalchol gel according to the labelling as well as known or suspected allergy to the specific product used in the study.
12. Contagious blood disease.
13. Known alcohol or drug abuse, or any condition associated with poor compliance.
14. Participation in a clinical study during the last 90 days before start of treatment.
15. Previous enrolment or randomisation in the present study -

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-01 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity, | q2 2007- q3 2008

SECONDARY OUTCOMES:
Glucose tolerance, HbA1c levels, Abdominal obesity, prostate safety, Sexual function, Sleepiness, Urinary symptoms, Hypogonadal symptoms score | Q 2 2007 - q 3 2008

CONTACTS AND LOCATIONS:
Overall Officials: Urban Ekström, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden